CLINICAL TRIAL: NCT05368896
Title: Peri-OPerative InflamMAGing in Elderly Patients Undergoing Major Surgery: Prediction and Pathomechanisms of Post-operative Morbidities
Brief Title: Peri-operative Inflammaging in the Elderly After Surgery
Acronym: POPIMAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. Christian Bode, Principal Investigator, University of Bonn
Other Study IDs: KAI-1
Record Dates: First submitted 2022-04-05; First posted 2022-05-10 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Aging; Immunology; Postoperative Complications; Surgery
Keywords: Frailty; Neuro-Degenerative Disease; innate immunity; immunphenotyping
MeSH Terms: conditions — Postoperative Complications; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients with postoperative complications after major surger: Patients >80 years that will undergo major visceral or orthopedic surgery

SUMMARY:
The population older than 80 years will significantly increase in the near future. Older patients' cognitive and physical status is known to deteriorate after surgery, leading to a high 30-day mortality due to post-operative comorbidities. Aging and related diseases share immune-related pathomechanisms. During aging, a chronic, low-grade sterile inflammation, called inflamaging, gradually develops. This likely results from low-grade innate immune activation and a functional, epigenomic and transcriptomic reprogramming of immune cells. Based on the hypothesis that surgical trauma leads to misplaced or altered self-molecules, which exacerbate inflammation and the postoperative risk for morbidity and mortality in elderly patients. There is increasing evidence that the individual's pre-operative immunobiography determines the susceptibility to peri-operative inflammation and post-operative outcome. Current exploratory pilot study will thus perform phenotyping of patients above 80 years undergoing major surgery. Participants will be evaluated for acute and long-term outcomes, including all-cause mortality, physical and cognitive function. To assess the individual's immunobiography, participants will be characterised by inflammation biomarkers combined with immunophenotyping, functional assays, and (epi-) genomic analyses before and after surgery. The cognitive impairment will be evaluated by measuring markers of neurodegeneration and neuropsychiatric testing and relate findings to volumetric imaging using high-resolution MRI to identify brain changes associated with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 80 years
* elective major surgery defined as knee / hip replacement, spondylodesis (> 2 levels), gastrectomy, resection of esophagus, liver, pancreas, colon, rectum or lung

Exclusion Criteria:

* no informed consent
* not able to perform neurocognitive testing
* preexisting infection systemic: CRP>100 mg/l, Leukos >12.0 G/l or clinical signs

Prosthetic joint infection (MSIS 2011 criteria):

PJI is present when 1 major criteria exist or 4 out of 6 minor criteria exist

Major criteria:

* 2 positive periprosthetic cultures with phenotypically identical organisms
* A sinus tract communicating with the joint

Minor criteria:

* Elevated CRP and ESR
* Elevated synovial fluid WBC count or ++ change on leukocyte esterase test strip
* Elevated synovial fluid PMN%
* Presence of purulence in the affected joint
* Positive histologic analysis of periprosthetic tissue
* A single positive culture
* Immunosuppression (HIV, glucocorticoids, immunosupressants)
* Autoimmune diseases
* ongoing or recent (<3 months) chemo/radiotherapy

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 80 years undergoing major surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Peri-interventional (surgical and non-surgical interventional) all-cause mortality rate on day 30 | 30 days
  Number of patients with death from any cause
In-hospital outcome according to the ACS National Surgical Quality Improvement Program® (ACS NSQIP®) | 30 days
  Number of patients with e.g. pneumonia, cardiovascular complication, surgical site infection, urinary tract infection, venous thromboembolism, acute or progressive renal failure and re-surgery

SECONDARY OUTCOMES:
Analysis of the new-onset of serious cardiac complications | 30 days
  Number of patients with serious cardiac complication
  Cardiac complication is defined according to the American Heart Association
Analysis of the new-onset of serious pulmonary complications | 30 days
  Number of patients with
  Pneumonia: Clinical or radiological diagnosis. or Pulmonary embolism: Radiological diagnosis. Signs of pneumonia or pulmonary embolism in the autopsy
Analysis of the new-onset of acute stroke | 30 days
  Number of patients with new-onset of acute stroke, defined as a new focal or generalised neurological deficit of >24h duration in motor, sensory, or coordination functions with compatible brain imaging and confirmed by a neurologist. Transient ischemic attack is not considered as acute stroke. Signs of stroke in the autopsy.
Analysis of the new-onset of acute kidney injury | 30 days
  Number of patients with new-onset of acute kidney injury, defined according to the AKIN classification as AKI stage ≥2.
  This means increase of creatinine >2-3x from baseline within the hospital stay. Or urine output less than 0.5 ml kg-1 per hour for more than 12 hours. Or signs of acute kidney injury in the autopsy.
Unplanned intensive care unit admission | 30 days
  Number of patients
Unplanned intubation after intervention | 30 days
  Number of patients
Analysis of the new-onset of sepsis | 30 days
  Number of patients diagnoses by SEPSIS-3 definition
Analysis of the new-onset surgical side infection | 30 days
  Number of patients
Ventilator dependency >48 h | 48 hours
  duration of mechanical ventilation
Analysis of the new-onset thrombosis | 30 days
  number of patients with (deep) vein thrombosis
all cause mortality | 12 month
  Number of patients with death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mark Coburn, Prof, Study Chair — mark.coburn@ukbonn.de
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided